CLINICAL TRIAL: NCT01114100
Title: The Effects of Treatment With Sertraline for Panic Disorder and/or Depression Driven Chest Pain and/or Palpitations in a Double Blind, Care as Usual and Placebo Controlled Study
Brief Title: The Effects of Treatment With Sertraline for Noncardiac Chest Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Pfizer, Prof dr A Honig
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MEC99-128
Record Dates: First submitted 2010-04-29; First posted 2010-04-30 (Estimated); Last update posted 2010-05-18 (Estimated); Status verified 2010-05

CONDITIONS: Panic Attacks; Chest Pain; Depression
Keywords: chest pain; panic attacks; palpitations; depression; panic disorder; depressive disorder; non cardiac chest pain
MeSH Terms: conditions — Panic Disorder; Chest Pain; Depression; Depressive Disorder | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- sertraline, panic education (Active Comparator): treatment with sertraline after panic education
  Interventions: Drug: sertraline
- placebo after panic education (Placebo Comparator): treatment with placebo after panic education
  Interventions: Drug: placebo
- care as usual (No Intervention): patient received no diagnosis an no panic education, they had a 24 weeks follow up with a visit at 12 weeks and 24 weeks to evaluate their complaints

INTERVENTIONS:
Drug: sertraline — starting dose 25 mg for 1 week, the increasing to 50 mg, after each visit evaluation whether dosage has to be increased to maximally 150 mg
  Other Names: sertraline, zoloft
  Arms: sertraline, panic education
Drug: placebo — patients received 1 pill, according to their complaints the number of pills was increased to maximally 3
  Arms: placebo after panic education

SUMMARY:
The purpose of this study is to determine whether care as usual or intervention (consisting of sertraline versus placebo), are effective in the treatment of panic disorder and/or depression driven noncardiac chest pain.

DETAILED DESCRIPTION:
Noncardiac chest pain remains an important problem in clinical cardiology. Often, panic disorder and/or depression are the underlying cause. However, this is largely underdiagnosed.

There are no clear existing treatment strategies/methods for this specific patient population.

In our double blind, placebo controlled care as usual versus sertraline study, we want to investigate whether intervention is more effective as care as usual for diminishing chest pain, and also if sertraline is more effective in this specific population compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* chest pain without a cardiac cause
* diagnosed with panic disorder and or depression according to Diagnostic and statistical Manual (DSM) IV criteria
* Living < 50 km from the hospital
* informed consent

Exclusion Criteria:

* other primary DSM IV diagnosis
* known sensitivity to sertraline
* using other anti-depressive agents
* not speaking dutch language
* living in a nursery home or having dementia
* other severe, acute or progressive disease, kidney or liver-function disturbances, pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2000-01; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
panic attacks | 24 weeks
  reduction of panic attacks by more than or equal to 50%
17 items Hamilton depression (HAMD) rating scale score | 24 weeks
  reduction of HAMD score of >50%

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS)reduction score | 24 weeks
  reduction in Hospital Anxiety and Depression Score
Clinical Global Impression (CGI) improvement | 24 weeks
  improvement in Clinical Global Impression Scale
EuroQol (EQ-5D)score | 24 weeks
  improvement of Quality of Life measured by the EuroQol
Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) score | 24 weeks
  improvement of Quality of Life measured by the SF 36
health care costs | 24 weeks
  decrease of health care costs using a diary for health costs

CONTACTS AND LOCATIONS:
Overall Officials: Adriaan Honig, Prof,MD,Phd, Study Chair — Now: St Lucas and Andreas Hospital, Amsterdam, Netherlands; Petra Kuijpers, MD, PhD, Principal Investigator — Maastricht University Medical Centre, Maastricht, the Netherlands
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands